CLINICAL TRIAL: NCT03178227
Title: Randomized Trial of a Photoaging Mirroring Intervention to Prevent Smoking in Secondary Schools in Brazil - Study Protocol
Brief Title: Smokerface Mirroring in Brazil RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Titus J. Brinker, Titus J. Brinker, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SmokerfaceMirrorBrazil
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention is a school-based intervention involving photoaging of the students selfies which takes 45 minutes total.
  Interventions: Behavioral: Photoaging Mirroring Intervention
- Control (No Intervention): No intervention.

INTERVENTIONS:
Behavioral: Photoaging Mirroring Intervention — Medical students perform "mirroring" with the pupils in the schools where they shoot selfies with tablets and photoage them to future non-smokers vs. future smokers.
  Arms: Intervention

SUMMARY:
Before February 2018 the baseline survey is conducted in about 60 class in Brazilian secondary schools. These classes are randomized to control and intervention group in a 1/1 manner. A few weeks thereafter medical students from the local medical school visit the schools and perform a smoking prevention intervention called "photoaging mirroring intervention" which takes about 45 minutes. One month and six months after the intervention the intervention group receives another anonymous questionnaire monitoring smoking status. The primary endpoint is the difference in the chance of smoking prevalence between the two groups.

DETAILED DESCRIPTION:
Before February 2018 the baseline survey is conducted in about 60 class in Brazilian secondary schools. These classes are randomized to control and intervention group in a 1/1 manner. A few weeks thereafter medical students from the local medical school visit the schools and perform a smoking prevention intervention called "photoaging mirroring intervention" which takes about 45 minutes. One month and six months after the intervention the intervention group receives another anonymous questionnaire monitoring smoking status. The primary endpoint is the difference in the chance of smoking prevalence between the two groups.

ELIGIBILITY:
Inclusion Criteria:

Visiting a Brazilian secondary school

Exclusion Criteria:

Not visiting a Brazilian secondary school

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The difference of prevalences after six months | six months
  The primary outcome is the difference of the smoking prevalence from baseline to six months follow-up between the two groups.

SECONDARY OUTCOMES:
The difference of prevalences after one month | 1 month
  The secondary outcome is the difference of the smoking prevalence from baseline to one month follow-up between the two groups.

CONTACTS AND LOCATIONS:
Locations (2):
- University of Itauna, Itaúna, Brazil
- Titus Brinker, Bünde, Germany

REFERENCES:
- [Derived] Faria BL, Brieske CM, Cosgarea I, Omlor AJ, Fries FN, de Faria COM, Lino HA, Oliveira ACC, Lisboa OC, Klode J, Schadendorf D, Bernardes-Souza B, Brinker TJ. A smoking prevention photoageing intervention for secondary schools in Brazil delivered by medical students: protocol for a randomised trial. BMJ Open. 2017 Dec 10;7(12):e018589. doi: 10.1136/bmjopen-2017-018589. PMID 29229659